CLINICAL TRIAL: NCT00927368
Title: Comparison Between Ultrasound Guided Femoral Nerve Block Versus Ultrasound Guided Femoral Nerve Block With the Use of Peripheral Nerve Stimulation for Patients Undergoing Total Knee Replacement.
Brief Title: Comparison of 3 Techniques for Ultrasound-guided Femoral Nerve Catheter Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ehab Farag, Principal Investigator, Outcomes Research Consortium
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09-340
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Total Knee Replacement Surgery
Keywords: TKA; total knee replacement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ultrasound guidance alone (Active Comparator): The Tuohy needle was inserted in out-plane approach. Needle placement was considered adequate when the tip was visualized beneath the fascia iliaca; the catheter was then introduced 5 cm beyond the needle tip. Electrical stimulation was not used.
  Interventions: Procedure: ultrasound guidance alone
- Ultrasound guidance needle stimulation (Active Comparator): For the ultrasound guidance and needle stimulation arm, the Tuohy needle was positioned with the tip beneath the fascia iliaca under ultrasound guidance. The needle tip was then adjusted as necessary to obtain a quadriceps muscle response with a stimulating current ≤0.5 mA (2 Hz, pulse width 0.1 msec). Subsequently, the catheter was threaded 5 cm beyond the needle tip without additional electrical stimulation
  Interventions: Procedure: ultrasound guidance and needle stimulation
- Ultrasound guidance+catheter stimulation (Active Comparator): For the ultrasound guidance and catheter stimulation group, the Tuohy needle was positioned with the tip beneath the fascia iliaca under ultrasound guidance. The needle tip was then adjusted as necessary to obtain a quadriceps muscle response with a stimulating current ≤0.5 mA. At that point, the peripheral nerve stimulator was then disconnected from the stimulating needle and connected to the proximal end of the catheter. The catheter was then advanced 5 cm past the needle tip. If the motor response disappeared during catheter advancement, the catheter was withdrawn slightly until the response returned. Needle orientation and catheter advancement were adjusted as necessary to elicit quadriceps contractions via the catheter with a stimulating current ≤0.5 mA.
  Interventions: Procedure: ultrasound guidance and catheter stimulation

INTERVENTIONS:
Procedure: ultrasound guidance alone — The Tuohy needle was inserted in out-plane approach. Needle placement was considered adequate when the tip was visualized beneath the fascia iliaca; the catheter was then introduced 5 cm beyond the needle tip. Electrical stimulation was not used.
  Arms: Ultrasound guidance alone
Procedure: ultrasound guidance and needle stimulation — For the ultrasound guidance and needle stimulation group, the Tuohy needle was positioned with the tip beneath the fascia iliaca under ultrasound guidance. The needle tip was then adjusted as necessary to obtain a quadriceps muscle response with a stimulating current ≤0.5 mA (2 Hz, pulse width 0.1 msec). Subsequently, the catheter was threaded 5 cm beyond the needle tip without additional electrical stimulation.
  Arms: Ultrasound guidance needle stimulation
Procedure: ultrasound guidance and catheter stimulation — The Tuohy needle was positioned with the tip beneath the fascia iliaca under ultrasound guidance. The needle tip was then adjusted as necessary to obtain a quadriceps muscle response with a stimulating current ≤0.5 mA. At that point, the peripheral nerve stimulator was then disconnected from the stimulating needle and connected to the proximal end of the catheter. The catheter was then advanced 5 cm past the needle tip. If the motor response disappeared during catheter advancement, the catheter was withdrawn slightly until the response returned. Needle orientation and catheter advancement were adjusted as necessary to elicit quadriceps contractions via the catheter with a stimulating current ≤0.5 mA.
  Arms: Ultrasound guidance+catheter stimulation

SUMMARY:
This is a randomized study which will compare three femoral nerve catheter insertion techniques. Subjects will be randomized into one of thee groups, Group 1: ultrasound guided femoral nerve catheter using a stimulation needle and stimulating catheter, .Group 2: ultrasound guided femoral nerve catheter using a stimulation needle, but non-stimulating catheter, or Group 3: ultrasound guided femoral nerve block without stimulation.

DETAILED DESCRIPTION:
This is a randomized study which will compare three femoral nerve catheter insertion techniques. Subjects will be randomized into one of thee groups, Group 1: ultrasound guided femoral nerve catheter using a stimulation needle and stimulating catheter, .Group 2: ultrasound guided femoral nerve catheter using a stimulation needle, but non-stimulating catheter, or Group 3: ultrasound guided femoral nerve block without stimulation.

* Pain Scores after surgery with be measured using the VAS (Visual Analogue Scale). Subjects will be asked to rate their pain on a scale of 1-10.
* Block Performance time is the time from starting the block (after prepping and draping) until catheter is placed.
* Opioid requirements will be measured as the total amount of opioids (converted to morphine sulfate equivalents) used both during surgery, and during the first 48 hours after surgery.
* Block failure rate will be calculated as the rate of cases that requires repeating the block after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old at time of surgery.
* Male or female patients undergoing total knee replacement under either general or neuraxial anesthesia (spinal or epidural). Intraoperative, patients will receive spinal anesthetics with 15 mg bupivacaine and 25mcg of fentanyl intrathecally.

Exclusion Criteria:

* Current or recent drug abuse (within past 6 months).
* Pregnancy.
* Patient refuses regional analgesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Farag, M.D., Principal Investigator — The Cleveland Clinic; Daniel I Sessler, M.D., Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Guidance Alone | Ultrasound Guidance Needle Stimulation | Ultrasound Guidance+Catheter Stimulation
Started | 153 | 157 | 143
Completed | 147 | 152 | 138
Not Completed | 6 | 5 | 5
Not completed — enrollment in another study | 1 | 1 | 2
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — equipment failure | 1 | 0 | 0
Not completed — ineligible post randomization | 0 | 3 | 1
Not completed — cancellation of surgery | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Guidance Alone | Ultrasound Guidance Needle Stimulation | Ultrasound Guidance+Catheter Stimulation | Total
Number analyzed (Participants) | 147 | 152 | 138 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9) | 61 (13) | 63 (9) | 62 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 76 | 236
  Male | 67 | 72 | 62 | 201

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Average Verbal Response Scale Pain Score
Description: Time weighted average of verbal response scale (VRS) pain score on a scale from 0 (no pain) to 10 (worst pain imaginable).
  Verbal Response Scale (VRS) pain scores after surgery - which ranged from 0 (no pain) to 10 (maximum intolerable pain) - were assessed every 30 minutes in the recovery area and every 4 hours thereafter up to 48 hours postoperatively. These individual measurements were averaged for each patient using a time-weighted formula. (For a given patient, the observed VRS pain score profile as a function of time was linearly interpolated and integrated using the trapezoidal rule; then, the time-weighted average was calculated as the value of this integral divided by the total monitoring time of 48 hours.).
Time Frame: 48 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultrasound Guidance Alone | Ultrasound Guidance Needle Stimulation | Ultrasound Guidance+Catheter Stimulation
Number analyzed (Participants) | 147 | 152 | 138
units on a scale | 3.52 (1.62) | 3.24 (1.55) | 3.40 (1.47)
Statistical Analysis 1: Comparison: Ultrasound Guidance Needle Stimulation vs Ultrasound Guidance+Catheter Stimulation; The primary analysis for pain was a linear regression model comparing stimulating needle to stimulating catheter on the mean time-weighted average pain score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — Noninferiority analysis used the 0.5-point noninferiority delta in a 1-tailed test of the treatment effect regression parameter (i.e., testing the null hypothesis that mean stimulating needle minus mean stimulating catheter is greater than 0.5 points); p < 0.001, t-test, 2 sided — Significance criterion of 0.00694 after adjusting for group sequential design and applying Holm Bonferroni procedure to account for multiple comparisons; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.61 to 0.29]
Statistical Analysis 2: Comparison: Ultrasound Guidance Needle Stimulation vs Ultrasound Guidance+Catheter Stimulation; The primary analysis for pain was a linear regression model comparing stimulating catheter to stimulating needle on the mean time-weighted average pain score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — Noninferiority analysis used the 0.5-point noninferiority delta in a 1-tailed test of the treatment effect regression parameter (i.e., testing the null hypothesis that mean stimulating catheter minus mean stimulating needle is greater than 0.5 points); p = 0.03, t-test, 2 sided — Significance criterion of 0.01735 after adjusting for group sequential design and applying Holm Bonferroni procedure to account for multiple comparisons; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.29 to 0.61]
Statistical Analysis 3: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance+Catheter Stimulation; The primary analysis for pain was a linear regression model comparing stimulating catheter to ultrasound alone on the mean time-weighted average pain score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — Noninferiority analysis used the 0.5-point noninferiority delta in a 1-tailed test of the treatment effect regression parameter (i.e., testing the null hypothesis that mean catheter minus mean ultrasound alone is greater than 0.5 points); p < 0.001, t-test, 2 sided — Significance criterion of 0.01041 after adjusting for group sequential design and applying Holm Bonferroni procedure to account for multiple comparisons; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.57 to 0.33]
Statistical Analysis 4: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance+Catheter Stimulation; The primary analysis for pain was a linear regression model comparing ultrasound alone to stimulating catheter on the mean time-weighted average pain score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — Noninferiority analysis used the 0.5-point noninferiority delta in a 1-tailed test of the treatment effect regression parameter (i.e., testing the null hypothesis that mean ultrasound alone minus mean catheter is greater than 0.5 points); p = 0.02, t-test, 2 sided — Significance criterion of 0.01388 after adjusting for group sequential design and applying Holm Bonferroni procedure to account for multiple comparisons; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.33 to 0.57]
Statistical Analysis 5: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance Needle Stimulation; The primary analysis for pain was a linear regression model comparing stimulating needle to ultrasound alone on the mean time-weighted average pain score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — Noninferiority analysis used the 0.5-point noninferiority delta in a 1-tailed test of the treatment effect regression parameter (i.e., testing the null hypothesis that mean stimulating needle minus mean ultrasound alone is greater than 0.5 points); p < 0.001, t-test, 2 sided — Significance criterion of 0.00347 after adjusting for group sequential design and applying Holm Bonferroni procedure to account for multiple comparisons; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.72 to 0.16]
Statistical Analysis 6: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance Needle Stimulation; The primary analysis for pain was a linear regression model comparing ultrasound alone to stimulating needle on the mean time-weighted average pain score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — Noninferiority analysis used the 0.5-point noninferiority delta in a 1-tailed test of the treatment effect regression parameter (i.e., testing the null hypothesis that mean ultrasound alone minus mean stimulating needle is greater than 0.5 points); p = 0.11, t-test, 2 sided — Significance criterion of 0.02082 after adjusting for group sequential design and applying Holm Bonferroni procedure to account for multiple comparisons; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.16 to 0.72]

2. Primary Outcome: Opioid Consumption
Description: cumulative opioid consumption, where all opioids were converted to IV morphine equivalents
Time Frame: 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | Ultrasound Guidance Alone | Ultrasound Guidance Needle Stimulation | Ultrasound Guidance+Catheter Stimulation
Number analyzed (Participants) | 147 | 152 | 138
mg morphine equivalents | 57 [40 to 81] | 58 [39 to 80] | 55 [38 to 85]
Statistical Analysis 1: Comparison: Ultrasound Guidance Needle Stimulation vs Ultrasound Guidance+Catheter Stimulation; The primary analysis for opioid was a linear regression model comparing stimulating catheter to stimulating needle on the log of cumulative opioid consumption score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.04, t-test, 2 sided — [p-value comment as in outcome 1, analysis 6]; Mean Difference (Final Values) = 5, 95% CI 2-sided [-17 to 34]
Statistical Analysis 2: Comparison: Ultrasound Guidance Needle Stimulation vs Ultrasound Guidance+Catheter Stimulation; The primary analysis for opioid was a linear regression model comparing stimulating needle to stimulating catheter on the log of cumulative opioid consumption score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.002, t-test, 2 sided — [p-value comment as in outcome 1, analysis 5]; Mean Difference (Final Values) = -5, 95% CI 2-sided [-25 to 21]
Statistical Analysis 3: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance+Catheter Stimulation; The primary analysis for opioid was a linear regression model comparing stimulating catheter to ultrasound alone on the log of cumulative opioid consumption score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — Noninferiority analysis used the 0.5-point noninferiority delta in a 1-tailed test of the treatment effect regression parameter (i.e., testing the null hypothesis that mean stimulating catheter minus mean ultrasound alone is greater than 0.5 points); p = 0.03, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 3, 95% CI 2-sided [-25 to 21]
Statistical Analysis 4: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance+Catheter Stimulation; The primary analysis for opioid was a linear regression model comparing ultrasound alone to stimulating catheter on the log of cumulative opioid consumption score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — Noninferiority analysis used the 0.5-point noninferiority delta in a 1-tailed test of the treatment effect regression parameter (i.e., testing the null hypothesis that mean ultrasound alone minus mean stimulating catheter is greater than 0.5 points); p = 0.005, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3, 95% CI 2-sided [-24 to 23]
Statistical Analysis 5: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance Needle Stimulation; The primary analysis for opioid was a linear regression model comparing stimulating needle to ultrasound alone on the log of cumulative opioid consumption score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 5]; p = 0.006, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = -2, 95% CI 2-sided [-22 to 25]
Statistical Analysis 6: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance Needle Stimulation; The primary analysis for opioid was a linear regression model comparing ultrasound alone to stimulating needle on the log of cumulative opioid consumption score for a patient in the first 48 hours; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 6]; p = 0.02, t-test, 2 sided — [p-value comment as in outcome 1, analysis 4]; Mean Difference (Final Values) = 2, 95% CI 2-sided [-20 to 29]

3. Secondary Outcome: Block Performance Time
Description: Block performance time, defined as the time from block start until catheter placement.
Time Frame: time elapsed from beginning the block to catheter placement
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Ultrasound Guidance Alone | Ultrasound Guidance Needle Stimulation | Ultrasound Guidance+Catheter Stimulation
Number analyzed (Participants) | 147 | 152 | 138
seconds | 110 [85 to 135] | 150 [126 to 175] | 177 [151 to 202]
Statistical Analysis 1: Comparison: Ultrasound Guidance Needle Stimulation vs Ultrasound Guidance+Catheter Stimulation; Stimulating needle versus stimulating catheter; Test type: Superiority or Other; p = 0.11, ANOVA
Statistical Analysis 2: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance Needle Stimulation; Stimulating needle versus ultrasound guidance alone; Test type: Superiority or Other; p = 0.01, ANOVA; Mean Difference (Final Values) = 40, 95% CI 2-sided [6 to 75]
Statistical Analysis 3: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance+Catheter Stimulation; Stimulating catheter versus ultrasound guidance alone; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 67, 95% CI 2-sided [31 to 102]

4. Secondary Outcome: Incremental Cost of Femoral Nerve Blocks
Description: The incremental cost between strategies was calculated as the additional cost of one strategy to the next less costly strategy. There was no variance in the price because these prices were contracted with the hospital. The contracted price for a hospital does not change or fluctuate.
Time Frame: postoperative period when block is used
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Ultrasound Guidance Alone | Ultrasound Guidance Needle Stimulation | Ultrasound Guidance+Catheter Stimulation
Number analyzed (Participants) | 153 | 157 | 143
dollars | 14 (0) | 36 (0) | 50 (0)
Statistical Analysis 1: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance Needle Stimulation; We calculated incremental cost, defined as the additional cost of one strategy to the next less costly strategy; Test type: Superiority or Other; incremental cost, measured in dollars = 14 — Incremental cost (additional cost of stimulating needle compared to ultrasound alone)
Statistical Analysis 2: Comparison: Ultrasound Guidance Needle Stimulation vs Ultrasound Guidance+Catheter Stimulation; We calculated incremental cost, defined as the additional cost of one strategy to the next less costly strategy; Test type: Superiority or Other; incremental cost, measured in dollars = 36 — We estimated incremental cost, or additional cost of stimulating needle + catheter stimulation to stimulating needle alone
Statistical Analysis 3: Comparison: Ultrasound Guidance Alone vs Ultrasound Guidance+Catheter Stimulation; We calculated incremental cost, defined as the additional cost of one strategy to the next less costly strategy; Test type: Superiority or Other; incremental cost, measured in dollars = 50 — We calculated incremental cost, or the additional cost of stimulating needle + stimulating catheter to ultrasound alone

ADVERSE EVENTS:
Arm/Group | Ultrasound Guidance Alone | Ultrasound Guidance Needle Stimulation | Ultrasound Guidance+Catheter Stimulation
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/152 | 0/138
Other Adverse Events (participants affected / at risk) | 0/147 | 0/152 | 0/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No